CLINICAL TRIAL: NCT07330388
Title: The Effects of Probiotics on Metabolic Biomarkers, Inflammation, and the Antioxidant System in Patients With Type 2 Diabetes Mellitus
Brief Title: Probiotic Effects in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Asli Kilavuz, Assoc. Prof., MD, PhD, Ege University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-4.1/67; TGA-2020-20200 (Other Grant/Funding Number: Ege University Scientific Research Projects Unit)
Record Dates: First submitted 2025-12-10; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Diabetes Mellitus (Type 2); Inflammation; Probiotics; Antioxidant Effect; Glucose Metabolism; Lipid Metabolism
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Inflammation

STUDY DESIGN:
Intervention Model Description: Participants were allocated sequentially according to order of presentation (alternate allocation). According to the order of presentation to the outpatient clinic, the first patient who met the inclusion criteria was included in the probiotic group and the second patient who presented to the outpatient clinic was included in the control group. Patients in the intervention group were given a probiotic supplement containing Lactobacillus acidophilus, Lactobacillus rhamnosus, Bifidobacterium lactis and Lactobacillus paracasei, each containing 1.25 billion live microorganisms, without vitamins and minerals, twice a day in addition to their current treatment for 12 weeks (Probiotic group). Patients in the control group were not given any additional treatment and were allowed to continue their antidiabetic treatment for 12 weeks (Control group).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic group (Experimental): Patients in the intervention group were given a probiotic supplement containing Lactobacillus acidophilus, Lactobacillus rhamnosus, Bifidobacterium lactis and Lactobacillus paracasei, each containing 1.25 billion live microorganisms, without vitamins and minerals, twice a day in addition to their current treatment for 12 weeks.
  Interventions: Dietary Supplement: Probiotic group
- Control group (No Intervention): Patients in the control group were not given any additional treatment and were allowed to continue their routine antidiabetic treatment for 12 weeks

INTERVENTIONS:
Dietary Supplement: Probiotic group — Patients in the intervention group were given a probiotic supplement containing Lactobacillus acidophilus, Lactobacillus rhamnosus, Bifidobacterium lactis and Lactobacillus paracasei, each containing 1.25 billion live microorganisms, without vitamins and minerals, twice a day in addition to their current treatment for 12 weeks (Probiotic group). Patients in the control group were not given any additional treatment and were allowed to continue their routine antidiabetic treatment for 12 weeks (Control group).
  Arms: Probiotic group

SUMMARY:
Adult-onset diabetes is a disease characterized by high blood glucose levels and is one of the leading causes of cardiovascular disease, blindness, end-stage renal failure, and hospitalization. Recent studies support the idea that bacteria found in the gut may play an important role in the development and progression of diabetes. Changes in the gut bacterial environment can affect blood glucose and blood lipids. A increasing number of recent studies have shown that probiotics can alter the gut bacterial environment and reduce blood glucose and blood lipids. The aim of this study is to investigate the effects of probiotics, administered in addition to your current medications, on blood glucose and blood lipids.

DETAILED DESCRIPTION:
Participants aged 35-65 years diagnosed with T2DM were allocated sequentially according to order of presentation to either probiotic group (n=39) or control group (n=38). The intervention group received a multi-strain probiotic supplement containing Lactobacillus acidophilus, Lactobacillus rhamnosus, Bifidobacterium lactis and Lactobacillus paracasei, twice daily for 12 weeks, while the control group continued standard care. This study evaluated anthropometric measurements, eating attitudes, dietary frequency, quality of life, and physical activity. Biochemical analyses included glycemic control, lipid profiles, inflammation markers (high-sensitivity C-Reactive Protein, Ceruloplasmin), and oxidative stress markers (Malondialdehyde, Glutathione).

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 35-65 years
* Previously diagnosed with T2DM
* Volunteering to participate in this study.

Exclusion Criteria:

* Use of any systemic antibiotics, multivitamins, minerals, herbal medicines, prebiotic, probiotic and postbiotic supplements in the last 3-6 months
* Having a diagnosis of any inflammatory bowel disease, severe renal dysfunction or hepatic dysfunction, immunodeficiency diseases, acute infection, rheumatoid arthritis, cancer history
* history of alcohol abuse or drug dependence,
* pregnant or lactating women

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Efficacy of probiotics on inflammatory markers | From enrollment to the end of treatment at 12 weeks
  hs-CRP
Efficacy of probiotics on inflammatory markers | From enrollment to the end of treatment at 12 weeks
  Ceruloplasmin
Efficacy of probiotics on antioxydant systems | From enrollment to the end of treatment at 12 weeks
  Glutathion
Efficacy of probiotics on antioxydant systems | From enrollment to the end of treatment at 12 weeks
  malondialdehyde

SECONDARY OUTCOMES:
Efficacy of probiotics on glucose metabolism | From enrollment to the end of treatment at 12 weeks
  Postprandial Blood Glucose
Efficacy of probiotics on glucose metabolism | From enrollment to the end of treatment at 12 weeks
  Fasting Blood Glucose
Efficacy of probiotics on glucose metabolism | From enrollment to the end of treatment at 12 weeks
  HbA1c
Efficacy of probiotics on lipid metabolism | From enrollment to the end of treatment at 12 weeks
  LDL Cholesterol
Efficacy of probiotics on lipid metabolism | From enrollment to the end of treatment at 12 weeks
  HDL Cholesterol
Efficacy of probiotics on lipid metabolism | From enrollment to the end of treatment at 12 weeks
  Triglyceride

CONTACTS AND LOCATIONS:
Overall Officials: İskender İnce, Assoc. Prof., Study Chair — Coordinator of Scientific Research Projects
Locations (1):
- Ege University Faculty of Medicine, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (3):
  • Study Protocol (2018-04-17): https://cdn.clinicaltrials.gov/large-docs/88/NCT07330388/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-17): https://cdn.clinicaltrials.gov/large-docs/88/NCT07330388/SAP_001.pdf
  • Informed Consent Form (2018-04-17): https://cdn.clinicaltrials.gov/large-docs/88/NCT07330388/ICF_002.pdf